CLINICAL TRIAL: NCT01206400
Title: Effect of Pioglitazone on Testosterone in Eugonadal Men With Type 2 Diabetes Mellitus - A Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Dr SRIDHAR, PGIMER
Organization: PIMERIndia (Unknown)
Other Study IDs: pioglitazonetestosterone
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2010-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: eugonadal, testosterone
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pioglitazone vs placebo: 15 patients in pioglitazone group and 15 in placebo group

SUMMARY:
To study the effects of pioglitazone on the steroidogenic enzyme axis in eugonadal men with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Several clinical studies demonstrated that pioglitazone not only improves insulin sensitivity but also decreases plasma androgen concentrations (DHEAS and androstenedione) in women with polycystic ovary syndrome (PCOS) . However the reduction in the androgen levels in PCOS is whether secondary to increase in the insulin sensitivity or due to direct effect of thiazolidinediones on steroidogenesis is not known.So far, two human studies have been conducted regarding the effects of rosiglitazone (a thiazolidinedione group of drug) on testosterone level, one in healthy individuals and another was in patients of type 2 diabetes with hypogonadism . But these studies gave equivocal results as the study population were different. Hence we plan to study the effects of pioglitazone on the steroidogenic enzyme axis in eugonadal men with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c level of 7.5% or less on stable dosages of sulphonylurea (glimepiride 1-6mg/day) and metformin (1-2g/day) for at least six weeks and BMI of 20-30 kg/m2.

Exclusion Criteria:

* hepatic impairment, coronary artery disease and or heart failure, renal failure, those who requires insulin therapy or HbA1c >7.5%, presence of macular edema and serum albumin <3gm/dL.

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: 30 eugonadal men with type 2 diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-12 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
pioglitazone effect on testosterone level | three months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Anil Bhansoli, MD.DM, Study Chair — PGIMER,Chandigarh
Locations (1):
- PGIMER, Chandigarh, Chandigarh, India

REFERENCES:
- [Background] Kapoor D, Channer KS, Jones TH. Rosiglitazone increases bioactive testosterone and reduces waist circumference in hypogonadal men with type 2 diabetes. Diab Vasc Dis Res. 2008 Jun;5(2):135-7. doi: 10.3132/dvdr.2008.022. PMID 18537102